CLINICAL TRIAL: NCT00799331
Title: An Exploratory Phase I, Single Centre, Double-Blind, Randomised, Placebo-Controlled, Parallel-Group Study to Assess the Pharmacokinetics of Increasing Oral Doses of AZD5985 in Healthy Male Volunteers
Brief Title: Exploratory Study to Assess the Pharmacokinetics of AZD5985
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Christer Hultquist, Medical Science Director, AstraZeneca R&D Lund, Sweden
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D2300C00001; EudraCt No. 2008-005121-11
Record Dates: First submitted 2008-11-21; First posted 2008-11-27 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): AZD5985
  Interventions: Drug: AZD5985
- B (Experimental): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AZD5985 — Oral suspension. Single oral doses of AZD5985 starting with 4 mg and subsequently with up to 3 dose escalations will be administered not exceeding AstraZeneca pre-defined upper exposure limits.
  Arms: A
Drug: placebo — Oral suspension.
  Arms: B

SUMMARY:
The aim of this exploratory study is to assess the pharmacokinetics of increasing oral doses of AZD5985 in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures.
* Healthy male subjects aged 18 to 45 years (inclusive).
* Have a body mass index (BMI) between 19 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg.
* Be non-smoker or ex-smoker who has stopped smoking (or using other nicotine products) for >6 months prior to study start.

Exclusion Criteria:

* History or presence of any clinically significant disease or disorder in the opinion of the investigator.
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs or ECG at baseline in the opinion of the investigator.
* Participation in another investigational drug study within 3 months before Visit 2 or participation in a method development study (no drug) 1 month prior to Visit 2

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
It is the objective of this exploratory study to assess pharmacokinetics of AZD5985 following administration of single increasing doses. The primary variable is plasma concentration of AZD5985. | Frequent sampling occasions during study days

CONTACTS AND LOCATIONS:
Overall Officials: Eva Pettersson, Study Director — AstraZeneca R&D, Lund, Sweden; Maura Fallon, Principal Investigator — Parexel, Berlin, Germany
Locations (1):
- Research Site, Berlin, Germany